CLINICAL TRIAL: NCT01056692
Title: A Phase II Study of oc000459 in Subjects With Allergic Asthma; a Randomised, Double Blind, Two Way Balanced Crossover Comparing oc000459 With Placebo
Brief Title: OC000459 Bronchial Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Collaborators: Medicines Evaluation Unit, Manchester, UK (Unknown); King's College Hospital NHS Trust (Other)
Responsible Party: Dr David Singh, Medicines Evaluation Unit, Manchester UK
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/004/05
Record Dates: First submitted 2009-12-21; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Bronchial Asthma
Keywords: Asthma; bronchial allergen challenge; sputum eosinophiilia
MeSH Terms: conditions — Asthma | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active compound (Active Comparator): OC000459 orally
  Interventions: Drug: OC000459
- Placebo (Placebo Comparator): Placebo given orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OC000459 — Capsules twice daily for 15 days
  Arms: Active compound
Drug: Placebo — Capsules twice daily for 15 days
  Arms: Placebo

SUMMARY:
OC0000459 reduces inflammation in the tissues in response to allergic stimuli in patients with asthma. This clinical trial, in mildly asthmatic patients, studies the effects of OC000459 and placebo on the asthmatic response to two known stimulants of the asthmatic response in the lungs, namely cat hair, pollen or house dust mite and methacholine.

ELIGIBILITY:
Inclusion Criteria:

* Known history of asthma (intermittent wheezing, cough, dyspnoea responsive to inhaled short acting beta agonists).
* FEV1 >65% of predicted on at least two occasions at screening.
* At the screening allergen challenge, a decrease in FEV1 of ≥20% in the early asthmatic reaction and of ≥15% in the LAR to allergen on 3 separate occasions between 3-10hrs post allergen, 2 of which must be consecutive.
* No steroid usage in the past 12 weeks.
* Testing positive to skin prick challenge with at least one of the following allergens: house dust mite, pollen or cat hair within the previous 12 months.
* Non smokers for a minimum of 6 months; less than 10 pack year history.

Exclusion Criteria:

* Respiratory tract pathology other than allergic asthma.
* Lower respiratory tract infection within 4 weeks prior to an allergen challenge.
* Receipt of prescribed or OTC medication other than paracetamol or short acting inhaled beta agonists within 14 days of screening or of the first day of each dosing period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02

PRIMARY OUTCOMES:
The primary endpoint is the diminution in the late asthmatic response to bronchial allergen challenge as measured by the AUC and the maximum of percentage reductions in FEV1 between 3 and 10 hours after allergen challenge. | Primary outcome is measured after 15 days of treatment with active or placebo

SECONDARY OUTCOMES:
Secondary biological activity endpoints include the diminution of the early asthmatic response to bronchial allergen challenge sputum eosinophilia, the methacholine PC20 after allergen challenge and exhaled NO pre- and post-allergen. | These measures are examined after 15 days of treatment with either active or placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Singh, MD, Principal Investigator — Medicines Evaluation Unit, Manchester, UK
Locations (2):
- United Kingdom (2):
  - King's College London School of Medicine, London, London
  - Medicines Evaluation Unit, Manchester, Manchester

REFERENCES:
- [Derived] Singh D, Cadden P, Hunter M, Pearce Collins L, Perkins M, Pettipher R, Townsend E, Vinall S, O'Connor B. Inhibition of the asthmatic allergen challenge response by the CRTH2 antagonist OC000459. Eur Respir J. 2013 Jan;41(1):46-52. doi: 10.1183/09031936.00092111. Epub 2012 Apr 10. PMID 22496329